CLINICAL TRIAL: NCT02812966
Title: Lutonix or Inpact for tHE tReatment Of fEmeropopliteal Stenosis - Drug Coated Balloon
Acronym: HEROES-DCB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: new FDA information regarding drug-coated balloons
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C5000163
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Results first posted 2024-07-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; drug coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lutonix Drug Coated Balloon (Active Comparator): Lutonix 035 Drug coated Balloon Percutaneous Transluminal Angioplasty Catheter
  Interventions: Device: Lutonix
- IN.PACT Drug Coated Balloon (Active Comparator): IN.PACT Admiral Paclitaxel-Coated Percutaneous Transluminal Angioplasty Balloon Catheter
  Interventions: Device: IN.PACT

INTERVENTIONS:
Device: Lutonix — Drug Coated Balloons
  Arms: Lutonix Drug Coated Balloon
Device: IN.PACT — Drug Coated Balloons
  Arms: IN.PACT Drug Coated Balloon

SUMMARY:
Investigators hypothesize in patients presenting with significant peripheral arterial disease with clinical indications for treatment with angioplasty, there will be a difference in 12 month patency between the subjects with Lutonix 035 Drug coated Balloon Percutaneous Transluminal Angioplasty Catheter and IN.PACT Admiral Paclitaxel-Coated Percutaneous Transluminal Angioplasty Balloon Catheter.

DETAILED DESCRIPTION:
Investigators hypothesize in patients presenting with significant peripheral arterial disease with clinical indications for treatment with angioplasty, there will be a difference in the 12 month patency (defined as peak systolic velocity ratio <=2.4 at 12 month follow-up visit with no target lesion revascularization or target lesion bypass) between the subjects with Lutonix 035 Drug coated Balloon Percutaneous Transluminal Angioplasty Catheter and IN.PACT Admiral Paclitaxel-Coated Percutaneous Transluminal Angioplasty Balloon Catheter. Investigators will also assess and compare target lesion revascularization rates, safety profiles, adverse events, healthcare costs, and healthcare utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is willing and able to provide informed consent, willing and agrees to comply with regular follow up visits, testing, medication regimen compliance any another treatments deemed necessary for treatment of vascular disease.
2. Male or non-pregnant female
3. Age greater >=18 years of age
4. Patients with moderate to severe claudication or ischemic rest pain as defined by Rutherford 2-4 class symptoms
5. >=1 tibial run-off vessel at baseline
6. Angiographic criteria

   * >=70% stenosis (via visual angiographic estimate in the superficial femoral artery and/or popliteal arteries as appropriate)
   * 4-7 mm vessel diameter
   * <=15 cm for planned treatment segment length.
   * Planned treatment segments are to no further proximal than 1 cm from the bifurcation of the common femoral artery and no further distal than the 1 cm above the tibioperoneal trunk.
   * Lesions treated within the target vessel are either De Novo lesions or not previously stented restenotic segments of the superficial femoral artery and/or popliteal artery that are greater than 90 days from prior angioplasty procedure
   * If the target vessel was previously stented the treated lesion must be at least 3 cm from the previously placed stent
   * Lesion must be able to be treated with either drug coated balloon device based on the sizes specifications of both devices
   * Successful, uncomplicated crossing must be possible within the treated lesion either with or without a crossing device
   * Inflow artery must be free from significant occlusive disease (< 50%) as confirmed by visual estimation by angiography otherwise the inflow artery must be treated beforehand.
   * At least 1 patent vessel outflow from the target vessel treated must be present by angiography

Exclusion Criteria:

1. Unable to meet clinical criteria to have peripheral angioplasty and follow-up treatment (lab values and pregnancy test)
2. Contra-indicated to either drug coated balloon
3. < 18 years of age at time of consent and/or index procedure
4. Pregnant or breastfeeding
5. In-stent restenosis within the target lesion
6. Previously stented target lesion/vessel.
7. Target lesion/vessel previously treated with drug-coated balloon <12 months prior to randomization/enrollment.
8. Perforated vessel as evidenced by extravasation of contrast media prior to consent or enrollment.
9. Presence of other hemodynamically significant outflow lesions in the target limb requiring intervention <=30 days of consent or randomization.
10. Presence of aneurysm in the target vessel.
11. Major amputation in the target limb.
12. Subjects who have undergone prior surgery of the superficial femoral artery/proximal popliteal artery in the target limb to treat atherosclerotic disease.
13. Use of atherectomy, laser or other debulking devices in the target limb superficial femoral artery/proximal popliteal artery during the index procedure.
14. Acute ischemia and/or acute thrombosis of the superficial femoral artery/proximal popliteal artery prior to consent or randomization.
15. Known hypersensitivity or contraindication to contrast dye that, in the opinion of the local investigator, cannot be adequately pre-medicated.
16. Known hypersensitivity/allergy to the investigational stent system or protocol related therapies.
17. On dialysis or on an immunosuppressant therapy.
18. Concomitant renal failure (including serum creatinine >2.0 mg/dL.)
19. Occurrence of myocardial infarction or cerebrovascular accident <=6 months prior to consent.
20. Platelet count <80,000 mm3 or >600,000 mm3 or history of bleeding diathesis.
21. Unstable angina pectoris at the time of consent or randomization.
22. Septicemia at the time of consent or randomization.
23. Moderate to severely calcified lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-04; Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaafer Golzar, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Edward Hospital, Naperville, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Prairie Education and Research Collaborative, Springfield, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lutonix Drug Coated Balloon | IN.PACT Drug Coated Balloon
Started | 18 | 17
Completed | 17 | 17
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lutonix Drug Coated Balloon | IN.PACT Drug Coated Balloon | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 9 | 9 | 18
Sex: Female, Male [Count of Participants; unit: Participants] — Population: No data received on 4 subjects in the Lutonix Drug Coated Balloon arm. No data received on 4 subjects in the IN.PACT Drug Coated Balloon arm.
  Participants
    number analyzed (Participants) | 14 | 13 | 27
    Female | 10 | 8 | 18
    Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Primary Patency (Peak Systolic Velocity Ratio<=2.4)
Description: Peak systolic velocity ratio <=2.4 (by duplex ultrasound scanning) with no target lesion revascularization or target lesion bypass
Time Frame: 12 months
Population: Data were not collected.
  Insufficient number of participants enrolled to perform data analysis prior to study closure. No data displayed because outcome measure had zero total participants analyzed.
Arm/Group | Lutonix Drug Coated Balloon | IN.PACT Drug Coated Balloon
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Target Lesion Revascularization Rate
Description: To examine, describe and compare/contrast within and between Drug Coated Balloon groups.
  1. Target lesion revascularization rate
  2. Safety event rate
  3. Healthcare utilization costs
Time Frame: 12 months
Population: Data were not collected.
  Insufficient number of participants enrolled to perform data analysis prior to study closure.
Arm/Group | Lutonix Drug Coated Balloon | IN.PACT Drug Coated Balloon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: In this study we will only be collecting Adverse Events (AEs) related to the procedure or device, unanticipated adverse device effects (UADE), and all Serious Adverse Events (SAEs) from the time of enrollment/randomization through study exit, up to 12 months.
Description: Participants asked when they came in if there was an adverse event
Arm/Group | Lutonix Drug Coated Balloon | IN.PACT Drug Coated Balloon
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lutonix Drug Coated Balloon (N=18) | IN.PACT Drug Coated Balloon (N=17)
subdural hematoma (Nervous system disorders) | 1 (1) | 0 (0) — Subject presented with neck pain, left arm weakness, and was diagnosed subdural hematoma attributed to a fall. Subject was hospitalized and underwent multiple surgeries. Subject developed seizures, pneumonia, and required mechanical ventilation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT02812966/Prot_SAP_000.pdf